CLINICAL TRIAL: NCT07229144
Title: An Open-Label, Phase 1b, Multiple Ascending Dose Study of OM336 in Participants With Active Sjogren's Disease or Idiopathic Inflammatory Myopathy
Brief Title: OM336 in Seropositive Autoimmune Diseases
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ouro Medicines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OM336-SAI-1002
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Sjogrens Disease; Idiopathic Inflammatory Myopathy (IIM)
Keywords: OM336; Ouro
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OM336 Dose Escalation (Experimental): Participants will receive OM336 via subcutaneous injection in ascending dose cohorts
  Interventions: Drug: OM336

INTERVENTIONS:
Drug: OM336 — OM336 is an engineered bispecific antibody directed against BCMA and CD3

SUMMARY:
An early-phase clinical trial evaluating the safety, tolerability, and pharmacokinetics of OM336 in adult participants with seropositive autoimmune diseases. OM336 is administered subcutaneously in ascending dose cohorts.

DETAILED DESCRIPTION:
An open-label, multicenter, multiple ascending dose study evaluating safety, tolerability, and PK/ADA profile of OM336 in seropositive autoimmune diseases. Exploratory assessments include clinical response and biomarkers.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of active seropositive autoimmune disease
* Relapsed/refractory after ≥2 prior/ongoing treatments
* Body weight ≥ 50 kg
* Willing to comply with and study requirements and procedures

Key Exclusion Criteria:

* Previous treatment with a BCMA-targeted therapy
* Clinically significant infection within 3 months of screening
* Major surgery within 3 months of screening or planned during the study
* Pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 12 weeks
  Incidence and severity of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Safety and Tolerability | 52 weeks
  Incidence and severity of treatment-emergent adverse events (TEAEs)
To assess the pharmacokinetics (PK) of OM336 | 12 weeks
  Serum concentrations of OM336
Detection of anti-drug antibodies | 12 weeks
  Detection of anti-drug antibodies

IPD SHARING:
Plan to Share IPD: No